CLINICAL TRIAL: NCT04854837
Title: Safety of Remdesivir Treatment in COVID-19 Patients Requiring Hemodialysis
Acronym: REM-HD
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Istvan Takacs, Head of department, Semmelweis University
Other Study IDs: REM-HD
Record Dates: First submitted 2021-04-21; First posted 2021-04-22 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Covid19; End Stage Renal Failure on Dialysis
Keywords: Remdesivir safety; COVID-19; Hemodialysis
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodialysed patients received remdesivir: Remdesivir: day-1: 200 mg intravenously; day 2-5: 100 mg intravenously
  Interventions: Drug: Remdesivir
- Hemodialysed patients not received remdesivir: Standard of care

INTERVENTIONS:
Drug: Remdesivir — Remdesivir treatment
  Groups: Hemodialysed patients received remdesivir

SUMMARY:
The FDA approved the antiviral drug remdesivir for use in adults for the treatment of COVID-19 requiring hospitalization.

There are only limited data about the safety of the drug in hemodialysed patents. Chronic kidney disease is a risk factor in COVID-19 for developing severe disease.

The aim of our investigation is to observe the safety of remdesivir among hemodialysed patients requiring hospitalization for COVID-19.

We are going to compare two group's data:

1. Hemodialysed COVID-19 patients requiring hospitalization because of pneumonia and need of oxygen supplementation, and admitted after 12/Apr/2021 - these patients received remdesivir.
2. Hemodialysed COVID-19 patients requiring hospitalization because of pneumonia and need of oxygen supplementation, and admitted before 12/Apr/2021 - these patients did not receive remdesivir.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 ys. of age
* Ability to understand and sign informed consent form
* End stage kidney disease of any cause, requiring hemodialysis
* COVID-19 disease (with at least one positive SARS-CoV-2 RT-PCR or COVID-19 antigene quick test)
* Radiologic evidence for pneumonia
* Need for oxygen supplemental oxygen

Exclusion Criteria:

* Hemodynamically unstable patients (systolic blood pressure <90Hgmm; heart rate>120/min)
* Significant liver enzyme elevation at screening (ASAT or ALAT >2.5×ULN)
* QTc > 470 msec at baseline ECG (Bazett formule)
* Need for mechanical ventilation or intensive care unit admission
* Limited life expectancy (<3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysed COVID-19 patients requiring hospitalization
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Adverse event frequency | 14 days after completion of treatment
  Number of adverse events occuring through the observational period

SECONDARY OUTCOMES:
Significant ASAT elevation | continuously, 14 days after completion of treatment
  Number of patients with significant (>2× ULN or >5× baseline) serum aspartate aminotransferase elevation
Significant ALAT elevation | continuously, 14 days after completion of treatment
  Number of patients with significant (>2× ULN or >5× baseline) serum alanin aminotransferase elevation
Significant ALP elevation | continuously, 14 days after completion of treatment
  Number of patients with significant (>2× ULN or >5× baseline) serum alkaline phosphatase elevation
Significant seBi elevation | continuously, 14 days after completion of treatment
  Number of patients with significant (>2× ULN or >5× baseline) serum total bilirubin elevation
Frequency of suspected drug-induced injury | continuously, 14 days after completion of treatment
  Number of patients with drug induced liver injury
QTc prolongation | continuously, 14 days after completion of treatment
  Change in corrected QTc interval measured on 12-lead ECG, corrected by Bazett's formule
Arrhythmia occurence | continuously, 14 days after completion of treatment
  Number of patients with clinically significant (judged by investigator) ECG abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University - Department of Internal Medicine and Oncology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No